CLINICAL TRIAL: NCT06481007
Title: Algerian Cholecystectomy Outcomes and Determinants Study
Brief Title: ALgerian Cholecystectomy Outcomes and Determinants Study (AL-CODS)
Acronym: AL-CODS
Status: Not yet recruiting | Type: Observational
Sponsor: University of Oran 1 (Other)
Responsible Party: Principal Investigator, Anisse Tidjane, Professor, University of Oran 1
Other Study IDs: Univ-2024-0017
Record Dates: First submitted 2024-06-22; First posted 2024-07-01 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Cholecystectomy; Adults; Gall Stone; Polyps; Pancreatitis Biliary; Gallbladder Dyskinesia; Cholecystitis
Keywords: Algeria; Cholecystectomy; mortality; morbidity; 30 days; determinants
MeSH Terms: conditions — Gallstones; Polyps; Biliary Dyskinesia; Cholecystitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cholecystectomy: patient opérated ( cholecystectomy) and responding to inclusion criteria

SUMMARY:
Cholecystectomy, the surgical removal of the gallbladder, is a common procedure performed to treat benign gallbladder diseases such as cholelithiasis (gallstones), cholecystitis (inflammation of the gallbladder), and biliary dyskinesia. While generally considered safe, this surgery can be associated with significant morbidity and mortality, particularly in certain populations or healthcare settings. Understanding these outcomes and the factors influencing them is crucial for improving patient care and surgical practices.

In Algeria, the healthcare landscape presents unique challenges and opportunities for evaluating surgical outcomes. Limited studies have specifically focused on the morbidity and mortality associated with cholecystectomy in this context. This study aims to fill that gap by providing comprehensive data on 30-day postoperative outcomes following cholecystectomy for benign gallbladder diseases in Algeria. Such data is essential for benchmarking current practices, identifying areas for improvement, and ultimately enhancing patient safety and surgical efficacy.

DETAILED DESCRIPTION:
This study seeks to bridge this knowledge gap by offering detailed data on 30-day postoperative outcomes after cholecystectomy for benign gallbladder diseases in Algeria. This information is crucial for benchmarking existing practices, pinpointing areas for enhancement, and ultimately improving patient safety and surgical effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older.
* Undergoing cholecystectomy.
* Surgery performed in public or private hospitals in Algeria.
* Surgery performed from January 1, 2025, to June 30, 2025.

Exclusion Criteria:

* Patients younger than 18 years.
* Patients refusing to participate.
* Cholecystectomy performed for Gallbladder cancer.
* Cholecystectomy performed outside the inclusion period.
* Cholecystectomies performed in conjunction with other major surgeries.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients aged 18 years and older who undergo cholecystectomy for benign gallbladder diseases in Algeria. This includes patients who have their gallbladders removed due to conditions such as gallstones, cholecystitis, biliary dyskinesia and any other benign pathology
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-02 (Estimated)

PRIMARY OUTCOMES:
Evaluate the 30-day mortality and morbidity | occuring in of before 30 day postopérative période.
  Evaluation of rate of mortality and morbidity at 30 day
factors associated with 30-day morbidity and mortality | occuring in of before 30 day postopérative période.
  determinants of the occurence of complications and mortality on or before 30 day in postopérative period

SECONDARY OUTCOMES:
estimate the incidence of incidental gallbladder cancer discovered during cholecystectomy in Algeria. | postoperative periode ( during or after surgical procedure)
estimate the incidence of bile duct injuries following cholecystectomy for benign diseases | occuring in of before 30 day postopérative periode.
assess surgical practices related to cholecystectomy in Algeria. | During surgical procedure ( Cholecystectomy)

IPD SHARING:
Plan to Share IPD: No
we are not going to share data , but the study will be published in an open acces journal.